CLINICAL TRIAL: NCT01326884
Title: ZLP Clinical Study
Brief Title: Zenith Low Profile AAA Endovascular Graft (ZLP) Clinical Study
Acronym: ZLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-004
Record Dates: First submitted 2011-03-21; First posted 2011-03-31 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Abdominal Aortic Aneurysm; Aorto-iliac Aneurysm; Iliac Aneurysm
Keywords: aortic aneurysm; iliac aneurysm; endovascular procedures
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm; Aortic Aneurysm

ARMS (1):
- 1 (Other): Endovascular Repair
  Interventions: Device: ZLP

INTERVENTIONS:
Device: ZLP — ZLP Graft

SUMMARY:
A prospective study conducted in Japan to collect confirmatory peri-operative and 30-day information on use of the Zenith LP AAA Graft.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic, aorto-iliac, and iliac aneurysms of appropriate size
* Vessels suitable for endovascular access and aneurysm repair

Exclusion Criteria:

* Less than 20 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Composite rate of adverse clinical/device events | During (day 1) and after implantation through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Fairman, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- Japan (2):
  - Nara Medical University, Nara
  - Jikei University Hospital, Tokyo